CLINICAL TRIAL: NCT05081804
Title: The Effect of Enhanced Recovery After Surgery (ERAS) for Cesarean Section on Neonatal Blood Glucose - A Randomized Equivalency Trial
Brief Title: The Effect of Enhanced Recovery After Surgery (ERAS) for Cesarean Section on Neonatal Blood Glucose
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Arizona (Other)
Collaborators: Nova Biomedical (Industry)
Responsible Party: Principal Investigator, Karen Lesser, Associate Professor of Obstetrics and Gynecology, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ERAS-CS
Record Dates: First submitted 2021-10-04; First posted 2021-10-18 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Enhanced Recovery After Surgery; Cesarean Section
Keywords: ERAS; Neonatal hypoglycemia

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: The providers taking care of the neonates will not know if the mother was randomized to receive the intervention (carbohydrate drink).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Non-diabetic Control (No Intervention): Patients without diabetes. No intervention will be administered - standard care.
- Non-diabetic CHO Drink (Experimental): Patients without diabetes. Commercially available preoperative carbohydrate drink will be administered two hours prior to cesarean section.
  Interventions: Dietary Supplement: Carbohydrate Preoperative Drink
- Diabetic Control (No Intervention): Patients with diabetes. No intervention will be administered - standard care.
- Diabetic CHO Drink (Experimental): Patients with diabetes. Commercially available preoperative carbohydrate drink will be administered two hours prior to cesarean section.
  Interventions: Dietary Supplement: Carbohydrate Preoperative Drink

INTERVENTIONS:
Dietary Supplement: Carbohydrate Preoperative Drink — Patients randomized to the intervention will drink the preoperative drink two hours prior to surgery
  Arms: Diabetic CHO Drink; Non-diabetic CHO Drink

SUMMARY:
Enhanced Recovery After Surgery (ERAS) is a set of evidence-based guidelines that may be used during perioperative care for cesarean section. While there is good evidence that following ERAS protocols benefits postoperative recovery, less is understood about the effect on the fetus and neonate. This will be a randomized equivalence trial to determine if drinking a carbohydrate rich drink prior to cesarean section has an effect on neonatal glucose.

DETAILED DESCRIPTION:
Cesarean section is one of the most common surgeries performed today with over one million performed in the United States annually. Enhanced Recovery After Surgery (ERAS) is a standardized set of guidelines which has been utilized in multiple surgical disciplines, including colorectal, urologic, gynecologic, and hepatobiliary surgery. ERAS guidelines are now being adopted for the obstetric population and provide evidence-based guidelines for perioperative care for cesarean delivery. Part of the preoperative ERAS pathway includes the recommendation for oral administration of a carbohydrate- containing fluid prior to surgery. A Cochrane review found that across several trials, carbohydrate loading was associated with favorable outcomes such as decreased time to passage of gas and reduction in length of hospital stay. Maternal outcomes are improved due to the decrease in insulin resistance that perioperative carbohydrate loading provides. During surgery, the body enters a catabolic state leading to insulin resistance that may delay recovery. Preoperative carbohydrate drinks have also been given to patients with diabetes, and although the decrease in insulin resistance is less certain, there seems to be less risk of postoperative hyperglycemia and the practice is considered safe but needing more study.

While it is clear that ERAS provides benefits to the mother, less is understood about the effects on the fetus and neonate. Fetal and neonatal glucose level is known to be strongly tied to the level of insulin resistance and glucose level in the mother, particularly in the immediate time period prior to birth. Neonatal hypoglycemia after delivery is an important determinate of health, as hypoglycemia has been linked to poor neurologic outcomes. Cesarean section is a known risk factor for neonatal hypoglycemia requiring IV dextrose with an odds ratio of 1.4. There are known risk factors for neonatal hypoglycemia, such as being the infant of a diabetic mother, preterm, weight <2500g, or >4500g, and poor feeding, however, the incidence of hypoglycemia in neonates with no clear risk factors is 5-15%. With health care systems adopting the ERAS protocol as part of the standardized guidelines for perioperative care, it will be important to understand the effect of carbohydrate loading on both maternal and neonatal glucose levels as well as other outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Women with term pregnancies
* Intact Amniotic membranes
* Not in labor
* Planned delivery by cesarean section
* Fluent in either English or Spanish

Exclusion Criteria:

* Less than 18 years old
* In labor
* Not fasted at least 8 hours
* Did not do glucose screening during pregnancy
* Fetal anomalies
* History of galactosemia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2021-10-20 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Neonatal glucose (mg/dl) | 60-120 minutes of life
  Neonatal glucose (mg/dl)

SECONDARY OUTCOMES:
Neonatal glucose 2 (mg/dl) | 24 hours of life
  Neonatal glucose 2 (mg/dl)

CONTACTS AND LOCATIONS:
Locations (1):
- Banner University Medicial Center, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bilku DK, Dennison AR, Hall TC, Metcalfe MS, Garcea G. Role of preoperative carbohydrate loading: a systematic review. Ann R Coll Surg Engl. 2014 Jan;96(1):15-22. doi: 10.1308/003588414X13824511650614. PMID 24417824
- [Background] Fay EE, Hitti JE, Delgado CM, Savitsky LM, Mills EB, Slater JL, Bollag LA. An enhanced recovery after surgery pathway for cesarean delivery decreases hospital stay and cost. Am J Obstet Gynecol. 2019 Oct;221(4):349.e1-349.e9. doi: 10.1016/j.ajog.2019.06.041. Epub 2019 Jun 22. PMID 31238038
- [Background] Ge LN, Wang L, Wang F. Effectiveness and Safety of Preoperative Oral Carbohydrates in Enhanced Recovery after Surgery Protocols for Patients with Diabetes Mellitus: A Systematic Review. Biomed Res Int. 2020 Feb 18;2020:5623596. doi: 10.1155/2020/5623596. eCollection 2020. PMID 32219135
- [Background] Harris DL, Weston PJ, Harding JE. Incidence of neonatal hypoglycemia in babies identified as at risk. J Pediatr. 2012 Nov;161(5):787-91. doi: 10.1016/j.jpeds.2012.05.022. Epub 2012 Jun 23. PMID 22727868
- [Background] Smith MD, McCall J, Plank L, Herbison GP, Soop M, Nygren J. Preoperative carbohydrate treatment for enhancing recovery after elective surgery. Cochrane Database Syst Rev. 2014 Aug 14;2014(8):CD009161. doi: 10.1002/14651858.CD009161.pub2. PMID 25121931
- [Background] Steenhagen E. Enhanced Recovery After Surgery: It's Time to Change Practice! Nutr Clin Pract. 2016 Feb;31(1):18-29. doi: 10.1177/0884533615622640. Epub 2015 Dec 24. PMID 26703956
- [Background] Turner D, Monthe-Dreze C, Cherkerzian S, Gregory K, Sen S. Maternal obesity and cesarean section delivery: additional risk factors for neonatal hypoglycemia? J Perinatol. 2019 Aug;39(8):1057-1064. doi: 10.1038/s41372-019-0404-z. Epub 2019 Jun 18. PMID 31213637
- [Background] Wilson RD, Caughey AB, Wood SL, Macones GA, Wrench IJ, Huang J, Norman M, Pettersson K, Fawcett WJ, Shalabi MM, Metcalfe A, Gramlich L, Nelson G. Guidelines for Antenatal and Preoperative care in Cesarean Delivery: Enhanced Recovery After Surgery Society Recommendations (Part 1). Am J Obstet Gynecol. 2018 Dec;219(6):523.e1-523.e15. doi: 10.1016/j.ajog.2018.09.015. Epub 2018 Sep 18. PMID 30240657